CLINICAL TRIAL: NCT00701389
Title: A Double-Blind, Randomized, Placebo-Controlled, 3-Period, Single Dose Crossover Study to Evaluate the Safety, Tolerability, and Blood Pressure Effect of an Oral Dose of Sumatriptan Alone and in Combination With MK0974 in Migraine Patients
Brief Title: Study to Evaluate the Safety, Tolerability, and Blood Pressure Effect of an Oral Dose of Sumatriptan Alone and in Combination With MK-0974 (Telcagepant) in Migraine Patients (0974-026)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0974-026; 2008_500
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Sequence 1: A→C→D→B (Experimental): Participants receive the following: Period 1: single oral dose of 100 mg sumatriptan/600 mg telcagepant (Treatment A); Period 2: single oral dose of sumatriptan placebo/600 mg telcagepant (Treatment C); Period 3: single oral dose of sumatriptan placebo/telcagepant placebo (Treatment D); Period 4: single oral dose of 100 mg sumatriptan/telcagepant placebo (Treatment B). Each dosing period is separated by a 5-day washout.
  Interventions: Drug: telcagepant potassium; Drug: sumatriptan; Drug: sumatriptan placebo; Drug: telcagepant potassium placebo
- Sequence 2: B→D→C→A (Experimental): Participants receive the following: Period 1: single oral dose of 100 mg sumatriptan/telcagepant placebo (Treatment B); Period 2: single oral dose of sumatriptan placebo/telcagepant placebo (Treatment D): Period 3: single oral dose of sumatriptan placebo/600 mg telcagepant (Treatment C); Period 4:single oral dose of 100 mg sumatriptan/600 mg telcagepant (Treatment A). Each dosing period is separated by a 5-day washout.
  Interventions: Drug: telcagepant potassium; Drug: sumatriptan; Drug: sumatriptan placebo; Drug: telcagepant potassium placebo
- Sequence 3: C→B→A→D (Experimental): Participants receive the following: Period 1 :single oral dose of sumatriptan placebo/600 mg telcagepant (Treatment C), Period 2: single oral dose of 100 mg sumatriptan/telcagepant placebo (Treatment B); Period 3: single oral dose of 100 mg sumatriptan/600 mg telcagepant (Treatment A): Period 4: single oral dose of sumatriptan placebo/telcagepant placebo (Treatment D). Each dosing period is separated by a 5-day washout.
  Interventions: Drug: telcagepant potassium; Drug: sumatriptan; Drug: sumatriptan placebo; Drug: telcagepant potassium placebo
- Sequence 4: D→A→B→C (Experimental): Participants receive the following: Period 1: single oral dose of sumatriptan placebo/telcagepant placebo (Treatment D), Period 2: single oral dose of 100 mg sumatriptan/600 mg telcagepant (Treament A); Period 3: single oral dose of 100 mg sumatriptan/telcagepant placebo (Treatment B); Period 4: single oral dose of sumatriptan placebo/600 mg telcagepant (Treatment C). Each dosing period is separated by a 5-day washout.
  Interventions: Drug: telcagepant potassium; Drug: sumatriptan; Drug: sumatriptan placebo; Drug: telcagepant potassium placebo

INTERVENTIONS:
Drug: telcagepant potassium — Single oral dose of 2 x 300 mg capsules.
Drug: sumatriptan — single oral dose of 100 mg sumatriptan
Drug: sumatriptan placebo — single oral dose
Drug: telcagepant potassium placebo — single oral dose of 2 MK-0974 placebo capsules

SUMMARY:
Study to understand the effects of migraine treatments on blood pressure in participants with migraine. The primary hypothesis is that the effect on semi-recumbent mean arterial pressure following the coadministration of telcagepant and sumatriptan is similar to that following administration of sumatriptan alone. That is, the true mean treatment difference (sumatriptan with telcagepant sumatriptan alone) in time-weighted mean arterial pressure for 2.5 hours following dosing is less than 5 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* History of migraine for longer than 6 months.
* Free from migraine 24 hours before each dosing.
* Judged to be in good health.
* Nonsmoker

Exclusion Criteria:

* Under age of legal consent.
* Legally or mentally incapacitated or has significant emotional problems.
* Taking any medications from about 2 weeks before the first dose of study medication.
* Has had surgery or donated blood or participated in another investigation study within 4 weeks prior to screening
* Currently a regular user of any illicit drugs or has a history of drug/alcohol abuse within about 2 years
* Consumes more than 6 caffeinated beverages per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-11-20 (Actual); Primary Completion 2008-04-10 (Actual); Study Completion 2008-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Depre M, Macleod C, Palcza J, Behm M, de Lepeleire I, Han T, Panebianco D, Smith W, Blanchard R, Chodakewitz J, Murphy M, de Hoon J. Lack of hemodynamic interaction between CGRP-receptor antagonist telcagepant (MK-0974) and sumatriptan: results from a randomized study in patients with migraine. Cephalalgia. 2013 Dec;33(16):1292-301. doi: 10.1177/0333102413494272. Epub 2013 Jun 24. PMID 23798725
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0974-026&kw=0974-026&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 2: B→D→C→A: Participants receive the following: Period 1:single oral dose of 100 mg sumatriptan/telcagepant placebo (Treatment B); Period 2: single oral dose of sumatriptan placebo/telcagepant placebo (Treatment D): Period 3: single oral dose of sumatriptan placebo/600 mg telcagepant (Treatment C); Period 4:single oral dose of 100 mg sumatriptan/600 mg telcagepant (Treatment A). Each dosing period is separated by a 5-day washout.
Period: Period 1
Arm/Group | Sequence 1: A→C→D→B | Sequence 2: B→D→C→A | Sequence 3: C→B→A→D | Sequence 4: D→A→B→C
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1: A→C→D→B | Sequence 2: B→D→C→A | Sequence 3: C→B→A→D | Sequence 4: D→A→B→C
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1: A→C→D→B | Sequence 2: B→D→C→A | Sequence 3: C→B→A→D | Sequence 4: D→A→B→C
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1: A→C→D→B | Sequence 2: B→D→C→A | Sequence 3: C→B→A→D | Sequence 4: D→A→B→C
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Participants: All participants enrolled in the study
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Full Range); unit: years] | 35.0 [21 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Mean Arterial Pressure (Sumatriptan With Telcagepant Versus Sumatriptan Alone)
Description: In each treatment period (1 through 4), duplicate readings of semi-recumbent blood pressure (BP) were completed using an automated blood pressure machine at predose, 30, 60, 90, 120, 150, 180, and 360 minutes postdose. Mean arterial pressure (MAP) was calculated as follows: MAP = Diastolic Blood Pressure (DBP) + (0.33 * Pulse Pressure [PP]) where PP = Systolic Blood Pressure [SBP] minus DBP. Only mean arterial pressure measurements up to and including 150 minutes postdose (including the predose measurement) were used to calculate the time-weighted averages. Time-weighted averages for each participant were obtained by calculating the area under the measurement-time curve of mean arterial pressure divided by the time period over which measurements were made (i.e. 150 minutes).
Time Frame: Predose up to 150 minutes postdose of each treatment period (up to 10 weeks)
Population: Participants who were administered sumatriptan with telcagepant or sumatriptan alone in either Periods 1, 2, 3, or 4 regardless of sequence and had evaluable blood pressure data obtained.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Groups:
- 100 mg Sumatriptan/600 mg Telcagepant: Participants who received single oral dose of 100 mg sumatriptan/600 mg telcagepant in either period 1, 2, 3 or 4 of the crossover
- 100 mg Sumatriptan/Telcagepant Placebo: Participants who received single oral dose of 100 mg sumatriptan/telcagepant placebo in either Period 1, 2, 3, or 4 of the crossover
Arm/Group | 100 mg Sumatriptan/600 mg Telcagepant | 100 mg Sumatriptan/Telcagepant Placebo
Number analyzed (Participants) | 24 | 22
mmHg | 89.0 [85.1 to 92.8] | 87.5 [83.6 to 91.4]
Statistical Analysis 1: Comparison: 100 mg Sumatriptan/600 mg Telcagepant vs 100 mg Sumatriptan/Telcagepant Placebo; 100 mg sumatriptan/600 mg telcagepant minus 100 mg sumatriptan/telcagepant placebo; Test type: Non-Inferiority or Equivalence — If the upper bound of the 90% CI is less than 5 mmHg, the primary hypothesis would be supported; Mixed Effect Model; Difference in Least Squares Means = 1.5, 90% CI 2-sided [0.0 to 3.0]

2. Secondary Outcome: Time-weighted Mean Arterial Pressure (Telcagepant Versus Placebo)
Description: as for outcome 1
Time Frame: Predose up to 150 minutes postdose of each treatment period (up to 10 weeks)
Population: Participants who were administered telcagepant or placebo in either Periods 1, 2, 3, or 4 regardless of sequence.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Groups:
- Sumatriptan Placebo/600 mg Telcagepant: Participants who received single oral dose of sumatriptan placebo/600 mg telcagepant in either period 1, 2, 3 or 4 of the crossover
- Sumatriptan Placebo/Telcagepant Placebo: Participants who received single oral dose of sumatriptan placebo/telcagepant placebo in either Period 1, 2, 3, or 4 of the crossover
Arm/Group | Sumatriptan Placebo/600 mg Telcagepant | Sumatriptan Placebo/Telcagepant Placebo
Number analyzed (Participants) | 24 | 24
mmHg | 84.7 [80.8 to 88.6] | 83.5 [79.6 to 87.3]
Statistical Analysis 1: Comparison: Sumatriptan Placebo/600 mg Telcagepant vs Sumatriptan Placebo/Telcagepant Placebo; sumatriptan placebo/600 mg telcagepant minus sumatriptan placebo/telcagepant placebo; Test type: Superiority or Other; Mixed Effect Model; Difference in Least Squares Means = 1.2, 90% CI 2-sided [-0.2 to 2.7]

3. Secondary Outcome: Number of Participants Who Experienced an Adverse Event During the Study
Description: Participants were assessed throughout the study for adverse events. An adverse event was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an adverse event.
Time Frame: up to 14 days after last dose of study drug (up to 10 weeks)
Population: All Patients as Treated defined as all participants who received at least one dose of the investigational drug. Adverse events were reported by study drug taken at the time of the event and not by randomly assigned sequence.
Measure: Number; unit: Participants
Groups:
- Sumatriptan Placebo/Telcagepant Placebo: Participants who received single oral dose of sumatriptan placebo/telcagepant placebo in either period 1, 2, 3 or 4 of the crossover
Arm/Group | 100 mg Sumatriptan/600 mg Telcagepant | 100 mg Sumatriptan/Telcagepant Placebo | Sumatriptan Placebo/600 mg Telcagepant | Sumatriptan Placebo/Telcagepant Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24
Participants | 9 | 12 | 8 | 10

4. Secondary Outcome: Number of Participants Who Were Discontinued From Any Study Period Due to an Adverse Event
Description: Participants were assessed throughout the study for adverse events. An adverse event was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an adverse event. The number of participants who were discontinued from the study due to adverse event was summarized.
Time Frame: up to 10 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Groups:
- Sumatriptan Placebo/600 mg Telcagepant: Participants who received single oral dose of generic placebo/600 mg telcagepant in either Period 1, 2, 3, or 4 in the crossover
- Sumatriptan Placebo/Telcagepant Placebo: Participants who received single oral dose of generic placebo/telcagepant placebo in either period 1, 2, 3 or 4 of the crossover
Arm/Group | 100 mg Sumatriptan/600 mg Telcagepant | 100 mg Sumatriptan/Telcagepant Placebo | Sumatriptan Placebo/600 mg Telcagepant | Sumatriptan Placebo/Telcagepant Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 14 days after last dose of study drug (up to 10 weeks)
Description: All Patients as Treated defined as all participants who received at least one dose of the investigational drug. Adverse events were reported by study drug taken at the time of the event and not by randomly assigned sequence.
Arm/Group | 100 mg Sumatriptan/600 mg Telcagepant | 100 mg Sumatriptan/Telcagepant Placebo | Sumatriptan Placebo/600 mg Telcagepant | Sumatriptan Placebo/Telcagepant Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 5/24 | 7/24 | 5/24 | 7/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg Sumatriptan/600 mg Telcagepant (N=24) | 100 mg Sumatriptan/Telcagepant Placebo (N=24) | Sumatriptan Placebo/600 mg Telcagepant (N=24) | Sumatriptan Placebo/Telcagepant Placebo (N=24)
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 1 | 1
Migraine (Nervous system disorders) | 3 | 4 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.